CLINICAL TRIAL: NCT03810508
Title: A Natural History Study of Charcot-Marie-Tooth 4J (CMT4J)
Acronym: CMT4J
Status: Terminated | Type: Observational
Why Stopped: Discontinued CMT4J development program
Sponsor: Neurogene Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CMT4J-100
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Charcot-Marie-Tooth Disease; Hereditary Motor and Sensory Neuropathy IV
Keywords: CMT4J
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Refsum Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will also have the opportunity to have biospecimens stored for up to 10 years for future exploratory analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Charcot-Marie-Tooth 4J (CMT4J) is a rare inherited peripheral neuropathy often characterized by rapidly progressive, asymmetrical upper and lower extremity weakness, muscle atrophy leading to loss of ambulation, respiratory compromise and premature death with no available treatment.

The purpose of this study is to investigate the clinical characteristics and natural clinical progression of symptoms in individuals with CMT4J. This natural history study is important to better understand disease course to be able to determine clinically meaningful outcome measures for use in future clinical trials.

DETAILED DESCRIPTION:
Charcot-Marie-Tooth (CMT) diseases are the most common inherited motor and sensory neuropathies, composed of a group of pathologically and genetically distinct subtypes ranging from slowly to rapidly progressive disease.

CMT4J is a rare subtype of CMT caused by mutations in the FIG4 gene. Pediatric-onset disease can often be characterized by rapid progression of muscle weakness and atrophy, culminating in loss of ambulation and respiratory compromise and premature death. Adult-onset CMT4J can present with a more variable disease course.

No prospective natural history study for CMT4J has been reported. This study aims to prospectively investigate the natural history of CMT4J, and concurrently to identify potential outcome measures that could be used in future clinical trials. No investigational product will be provided in the study.

ELIGIBILITY:
Subjects must have a prior confirmed molecular (genetic) diagnosis of CMT4J by clinical presentation and genetic testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of CMT4J based on clinical presentation and genetic testing (known or suspected pathogenic mutation in FIG4).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Charcot Marie-Tooth Pediatric Scale (CMTPedS) | Change is being assessed from baseline measures every 6 months for up to five years
  This an 11 item scale is used in patients younger than 18 yrs of age and generates a linear score of disability.
Charcot-Marie-Tooth Neuropathy Score second version (CMTNSv2) | Change is being assessed from baseline measures every 6 months for up to five years
  This is a 36 point scale that monitors disease impairment and progression with a higher score signifies increased disability.
Charcot Marie-Tooth Functional Outcome Measure (CMT-FOM) | Change is being assessed from baseline measures every 6 months for up to five years
  This is a performance-based outcome assessment which measures limitations in functional abilities in adults.
CMT Health Index (CMTHI) | Change is being assessed from baseline measures every 6 months for up to five years
  The CMTHI is a disease-specific, adult patient reported outcome measure designed to capture the disease burden of inherited neuropathies in the context of a clinical trial.
Magnetic Resonance Imaging (MRI) of the calf muscles without contrast | Change is being assessed from baseline measures every 6 months for up to five years
  MRI of bilateral thigh and calf muscles will be performed to characterize the pattern of muscle involvement and evaluate the muscle fat fraction (MFF).
Nerve Conduction Study (NCS) | Change is being assessed from baseline measures every 6 months for up to five years
  NCS is an electrophysiological test to evaluate the sensory and motor responses in the upper and lower extremities.
Pulmonary Function Test, sitting and lying (PFT) | Change is being assessed from baseline measures every 12 months for up to five years
  The purpose of the PFT is to identify the severity and progression of pulmonary impairment, and will be performed every 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Beausoleil, Study Director — Neurogene Inc.
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No